CLINICAL TRIAL: NCT02929628
Title: Evaluate the Safety and Effectiveness Between Various Frequency Stimulation and Traditional High Frequency Stimulation for the Treatment of Patients With Parkinson's Disease
Brief Title: Evaluate the Safety and Effectiveness of Various Frequency Stimulation for Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-020
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with Various Frequency Stimulation (Experimental): Patients are in the condition of Various Frequency Stimulation
  Interventions: Device: Beijing PINS Programming
- Patients With Traditional Frequency Stimulation (Sham Comparator): Patients in the condition of Sham Comparator are Traditional Frequency Stimulation
  Interventions: Device: Beijing PINS Programming

INTERVENTIONS:
Device: Beijing PINS Programming — Using the programming control the Stimulator to change the parameter

SUMMARY:
Patients with an implantable electrical nerve stimulation system Patient criteria included: over 18 years of age,MMSE≥ 24 score; H-Y stage in medicine off condition>2.0;an ability to walk at least 10 meters independently;subscore≥2 for UPDRS part II item 15;subscore >1 for UPDRS part II item 14; permissions given by informed consent. Patients with serious diseases such as tumor, sever liver or kidney dysfunction were not selected in the clinical trials. Subjects participating in other clinical trials related or not related to these trials were not chosen.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age,male or female patients
* idiopathic Parkinson's disease
* had deep brain stimulaton implant
* H-Y>2.0 in the absence of L-dopa
* UPDRSII-14 item ≥1
* UPDRSII-15 item ≥2
* an ability to walk at least 10 meters independently

Exclusion Criteria:

* Patients with serious diseases such as tumor, sever liver or kidney dysfunction were not selected in the clinical trials
* epilepsy
* Pregnant female
* History of severe neuropsychiatric disease
* Patients are taking part in other clinical trials in recent several months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Changs in the score of Stand-Walk-Sit Test | 1、3、6 and 12 month

SECONDARY OUTCOMES:
Change of the score in UPDRS | 1,3,6,12 months of Various Frequency Stimulation
Change of the score in PDQ-39 | 1、3、6、12 months of Various Frequency Stimulation
Change of the score in the FOG-Q | 1、3、6、12 month of Various Frequency Stimulation

IPD SHARING:
Plan to Share IPD: Yes